CLINICAL TRIAL: NCT01778218
Title: A Single Center Pilot Study to Establish the 99mTc-EC-DG Imaging Protocol to Evaluate the Presence and Severity of Coronary Artery Disease
Brief Title: A Single Center Study to Establish the Imaging Protocol of 99mTc-EC-DG in Evaluating the Presence and Severity of Coronary Artery Disease (CAD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cell>Point LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CP-ECDG-C2
Record Dates: First submitted 2013-01-22; First posted 2013-01-29 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; CAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 99mTc-EC-DG (Experimental): 99mTc-EC-DG injection followed by SPECT imaging during a cardiac rest study (Visit 1) and an exercise/regadenoson study (Visit 2)
  Interventions: Radiation: Radiolabeled (99Tc) EC-DG (ethylenedicysteine-deoxyglucose

INTERVENTIONS:
Radiation: Radiolabeled (99Tc) EC-DG (ethylenedicysteine-deoxyglucose — An injection of Technetium ethylenedicysteine-deoxyglucose (99mTc-EC-DG) to yield a target activity of 25 mCi (range of 10-25 mCi) with no more than 250 micrograms of EC-DG to be administered (there must be a minimum of 24 hours between Visit 1 and 2 administrations). Investigational Product to be given by IV push.

SUMMARY:
This study will assess the safety and tolerability of the investigational radiolabeled imaging agent technetium-99m-labeled ethylenedicysteine-deoxyglucose (99mTc-EC-DG). Additionally, the study will determine the specific times to best image the heart using a SPECT camera with the investigational imaging agent and compare the images to those taken while undergoing the standard rest and exercise/regadenoson testing previously performed to detect the presence and severity of Coronary Artery Disease (CAD).

DETAILED DESCRIPTION:
The study will assess the safety and tolerability of technetium-99m-labeled ethylenedicysteine-deoxyglucose (99mTc-EC-DG).

An outcome will be to develop an imaging protocol for a multicenter trial that will measure the specific imaging parameters required for determination of sensitivity and specificity of 99mTc-EC-DG in a cardiovascular single photon emission computed tomography (SPECT) study compared to an exercise/regadenoson 99mTc- Sestamibi (MIBI) study for detection of the presence and, when available, severity of coronary artery disease (CAD) as documented by coronary angiography when available.

This study will be a single-center, prospective, open-label study of up to 6 patients with positive findings from a MIBI (99mTc-sestamibi) exercise/regadenoson study within 30 days for evaluation of CAD. Patients who meet study eligibility criteria will undergo a 99mTc-EC-DG rest study and a 99mTc-EC-DG exercise/regadenoson study. When possible, patients enrolled will have clinical plans for a coronary angiography study to confirm presence and severity of CAD.

This study will enroll up to 6 patients with a reversible perfusion defect indicative of CAD on a MIBI exercise/regadenoson study. These patients will undergo a 99mTc-EC-DG rest study and an exercise/regadenoson study.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Reversible perfusion defect indicative of CAD on a MIBI exercise/regadenoson study completed within 30 days prior to screening;
3. When possible, a coronary angiography will be clinically planned; patient and treating physician must be agreeable to completing the angiogram after the 99mTc-EC-DG exercise/regadenoson study in order for the procedure to be performed.
4. The patient is able to provide written informed consent to participate in this study

Exclusion Criteria:

1. Known cardiomyopathy or history of congestive heart failure (CHF) due to left ventricular systolic dysfunction (ejection fraction < 40%)
2. A scheduled coronary angiogram that prevents the 99mTc-EC-DG exercise/regadenoson or rest study visits from being completed prior to the angiogram
3. Plans to begin new anti-anginal therapy prior to completing the 99mTc-EC-DG rest/stress study visits
4. Contraindication for provocative stress testing based on American College of Cardiology/American Heart Association (ACC/AHA) guidelines for exercise or pharmacologic testing
5. Intolerance or inability to receive sestamibi or regadenoson, or an inability or unwillingness to exercise on a graded treadmill or receive pharmacologic stress
6. Inability to lie still for 30 minutes during image acquisition
7. Women of childbearing potential, unless willing to use adequate contraception throughout the duration of the trial. Adequate contraception is considered hormonal contraception for >3 months prior to entry, intrauterine device (IUD) in place for at least 3 months, double barrier methods (condoms, diaphragm or spermicide), or a partner with non-reversed vasectomy > 40 days prior to entry.
8. Pregnant (positive human chorionic gonadotropin [hCG]) pregnancy test at screening for women of childbearing potential) or nursing
9. History of malignant disease (excluding treated basal cell or squamous cell carcinoma of skin, or low grade cancers that are stable and do not interfere with exercise which may be allowed with permission from the Medical Monitor) within 5 years prior to screening. Resolution of a prior malignancy more than 5 years prior to screening must be deemed as cured by the Investigator
10. Any physical, psychological or substance abuse (drug or alcohol) condition which, in the opinion of the Investigator, would interfere with the ability to provide informed consent or comply with study instructions or may adversely affect the safety of the patient if enrolled in this trial
11. A known allergy to 99mTc-EC-DG or its components
12. Inability to adhere to requirements specific to the study site's protocols for imaging and exercise/pharmacological stress testing, including but not limited to, dietary restrictions and prohibited medications
13. Received an investigational drug within 30 days prior to this study
14. Enrolled in or plans to enroll in another clinical trial during this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety: The number of participants with Adverse Events | From screening through 7 days after Investigational Product administration

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bateman, MD, Principal Investigator — Cardiovascular Imaging Technologies
Locations (1):
- Cardiovascular Imaging Technologies, Kansas City, Kansas, United States

REFERENCES:
- See also: Sponsor Link — http://cellpointweb.com